CLINICAL TRIAL: NCT02714361
Title: A Double Blind Randomised Controlled Trial to Investigate the Effect of Vitamin D3 Supplementation on Iron Absorption and Hepcidin Response in Marginally Deficient and Iron Deficient Women
Brief Title: A Study to Investigate the Effect of Vitamin D3 Supplementation on Iron Status in Iron Deficient Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chester (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1078/15/SF/CSN
Record Dates: First submitted 2015-11-13; First posted 2016-03-21 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Iron Deficiency; Anemia; Deficiency, Nutritional, With Poor Iron Absorption; Vitamin D Deficiency
Keywords: Iron deficiency; Vitamin D; Iron absorption; Hepcidin
MeSH Terms: conditions — Iron Deficiencies; Anemia; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D3 supplement (Active Comparator): Participants will be asked to take 1 capsule of vitamin D3 supplement (1500 IU) (37.5ug) daily for a total duration of 8 weeks.
  Interventions: Dietary Supplement: Vitamin D3 supplement
- Placebo (Placebo Comparator): Participants will be asked to take 1 capsule of placebo (65% olive oil) daily for a total duration of 8 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 supplement — 1500 IU (37.5 mcg) Vitamin D3 capsules daily over 8 weeks (56 days)
  Other Names: Cholecalciferol
  Arms: Vitamin D3 supplement
Other: Placebo — 65% olive oil capsules daily over 8 weeks (56 days)
  Other Names: Non active ingredient
  Arms: Placebo

SUMMARY:
Iron is one of the most vital elements in humans as it plays a role in physiological functions such as transferring and storing oxygen, transporting electrons and catalysing numerous reactions, from oxidative metabolism to cellular proliferation. Iron deficiency can be attributed to poor absorption that leads to insufficient iron to meet body requirements. Oral iron supplements have been extensively used to treat iron deficiency and iron deficiency anaemia. However, the use of iron compounds in fortifying foods is one of the best practical approach to combat iron deficiency, while improving diet and food pattern involves long-term goal which can be challenging. Vitamin D has recently been shown to affect hepcidin levels, which in turn has effects on iron status but there are a limited number of studies investigating the hepcidin profile in humans following iron supplementation, and few data are available, especially in humans, despite its role as a primary iron absorption and homeostasis regulator. Although several studies have been carried out using iron fortified products, there is limited data on the potential effect of vitamin D on iron metabolism amongst iron deficient women in particular. Therefore, the present study aims to investigate the effect of vitamin D3 supplementation (1500 IU) consumed with iron fortified breakfast cereals on haematological indicators and hepcidin response in iron deficient women.

DETAILED DESCRIPTION:
Recruitment And Sampling Strategy :

Participants will be recruited within the University of Chester, UK only. Emails and posters/leaflets will be used as a medium of advertisement to the target group (staff and students). A total of 62 pre-menopausal women aged between 19 to 40 years old will be included in the study based on criteria described below. Eligibility will be based upon serum ferritin and also vitamin D concentrations at screening before the start of the study. Participants will be required to complete a screening questionnaire which will provide information about participant's health status, drugs/medication/supplement usage, and recent occurrences of illness/trauma/injury. A 6 ml venous blood will be drawn to assess concentrations of plasma ferritin vitamin D, haemoglobin and full blood counts, Participants with plasma ferritin concentrations below 20.0 µg/L and vitamin D concentration below 250 nmol/l will be included in the study. If the levels of haemoglobin are found to be in severe stage of anaemia, the potential participant will be notified and advised to consult their General Practitioner (GP) (haemoglobin levels < 8.0 g/dL). All eligible participants will be briefed on the study protocol before the beginning of the study, and the eligible participants will be given a Participant Information Sheet (PIS) and asked to provide written informed consent.

An 8 week, double blind, randomised controlled trial will be carried out in Chester, United Kingdom (UK). The 8 week intervention period was selected since more than 1 month is appropriate to generally enlarge the erythropoietic marrow and observe changes in red blood cell indices, especially in non-anaemic groups. Most vitamin D studies have used a supplement concentration of 1000 IU and reported no adverse effects in the participants. Some studies have used higher doses of 1600 or 4000 IU with no reported adverse outcomes in the participants.

Participants will be randomly allocated to 2 groups:

1. Fe group (iron fortified breakfast cereals and placebo)
2. Vitamin D group (iron fortified breakfast cereals and vitamin D3).

Each participant will consume 60 grams of iron fortified breakfast cereals containing a total of 9 mg of iron daily for 8 weeks with either vitamin D3 placebo or vitamin D3 (1500 IU) according to their assigned group. The participants will consume the iron fortified breakfast cereals in the morning, with 200 ml of semi-skimmed milk daily for a period of 8 weeks. The participants will consume the vitamin D or placebo in the evening with 200 ml of water. Participants will be asked to maintain their dietary habits and physical activity during the course of study. Participants will also be asked not to donate blood during the course of the study. The remaining supplements will be returned at the final clinic (week 8), and compliance will be estimated.

Participants will be required to attend 3 clinics in total over a period of 8 weeks, and they will be assessed at baseline (Day 0), interim (Week 4) and post intervention (Week 8). Participants will be requested to fast overnight for approximately 8 hours before all clinics. At each clinic, a 30 ml blood sample will be taken and both height (cm) and weight (kg) will be measured. Before the start and the end of the study, participants will be required to keep a 3-day food diary which includes 2 weekdays and 1 weekend day to represent the habitual dietary intake of the participant. Blood samples will be batch analysed at the end of the intervention to assess all biomarkers of iron status and vitamin D metabolism.

Sample size and justification :

Sample size was estimated using iron supplementation data from a study carried out by Scholz-Ahrens et al. (2004) in which a serum ferritin concentration post intervention at 8 weeks (mean ± S.D) of 17.7 ± 11.8 ug/l (Fe fortified milk group) and 10.6 ± 8.1 ug/l (non fortified milk group) was reported. With an effect size of 0.7015447, the total sample size required for each group in the proposed study is 26. Taking into account a 20% drop out rate, the total sample size required is 31 (Power = 0.80). Therefore, the total sample size needed for the whole study is 62. Sample size was estimated using of G Power Software Version 3.1.7.

Statistical Analysis:

All statistical analyses will be conducted with International Business Machines (IBM) Statistical Package for the Social Sciences (SPSS) Statistic Data Editor Software (Version 21). Assuming that the data is normally distributed after performing a Shapiro Wilks normality test, one-way analysis of variance (ANOVA) with repeated measures will be conducted to compare the mean differences for all measured parameters within each group at baseline, interim and post intervention. The changes in the measured parameters between the periods of the study will be analysed using paired t-test. Pearson's correlation test will be performed to investigate the relationship between hepcidin profile and iron status biomarkers. A non-parametric approach will be adopted if the data is not normally distributed for all analyses. Differences will be considered significant with a p value ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* women;
* aged 19-49 years;
* healthy;
* non-pregnant nor lactating;
* serum ferritin levels less than 20 ug/l and vitamin D concentration below 250 nmol/l.

Exclusion Criteria:

* history of gastrointestinal and metabolic disorders;
* have donated blood in the past 6 months;
* regularly consuming nutritional supplements;
* haemoglobin levels less than 8.0 g/dL.

Ages: 19 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in Ferritin Concentration from Baseline to 8 weeks | 0 and 8 weeks
  Blood biomarker of iron stores measured in plasma samples by Mini Vidas Biomerieux

SECONDARY OUTCOMES:
Change in Haemoglobin Concentration from Baseline to 8 weeks | 0,4,8 weeks
  Iron status biomarker measured in whole blood by Beckman Coulter haematological analyser
Change in Hepcidin Concentration from Baseline to 8 weeks | 0,4,8 weeks
  Iron metabolism biomarker measured in plasma samples by ELISA commercial kit
Change in Vitamin D Concentration from Baseline to 8 weeks | 0,4,8 weeks
  Vitamin D3 status measured in plasma samples by Mini Vidas Biomerieux
Change in Full Blood Count Concentration from Baseline to 8 weeks | 0,4,8 weeks
  Iron status biomarker measured in whole blood samples by Beckman Coulter haematological analyser
Change in Parathyroid Hormone (PTH) Concentration from Baseline to 8 weeks | 0,4,8 weeks
  Vitamin D metabolism biomarker in plasma samples measured by ELISA commercial kit
Change in Vitamin D Receptor (VDR) Concentration from Baseline to 8 weeks | 0,4,8 weeks
  Vitamin D metabolism biomarker measured in plasma samples by ELISA commercial kit
Change in Calcium Concentration from Baseline to 8 weeks | 0,4,8 weeks
  Vitamin D metabolism biomarker measured in plasma samples by ELISA commercial kit
Change in Calcitriol Concentration from Baseline to 8 weeks | 0,4,8 weeks
  Vitamin D metabolism biomarker measured in plasma samples by ELISA commercial kit
Change in Ferritin Concentration from Baseline to 8 weeks | 0,4,8 weeks
  Iron status biomarker measured in plasma samples by Mini Vidas Biomerieux

CONTACTS AND LOCATIONS:
Overall Officials: Sohail Mushtaq, PhD, Principal Investigator — University of Chester
Locations (1):
- University of Chester, Chester, Cheshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The results are in the writing phase, and will be available in thesis form and possibly publication. It will be available in thesis form in 2017 and publication expected to be in 2018.

REFERENCES:
- [Background] Ahmad Fuzi SF, Mushtaq S. Vitamin D3 supplementation for 8 weeks leads to improved haematological status following the consumption of an iron-fortified breakfast cereal: a double-blind randomised controlled trial in iron-deficient women. Br J Nutr. 2019 May;121(10):1146-1157. doi: 10.1017/S0007114519000412. Epub 2019 Mar 1. PMID 30819262